CLINICAL TRIAL: NCT03926260
Title: Non-controlled Prospective Pilot Study Assessing Prognostic Performance of Circulating Tumour DNA Kinetic Analysis for Monitoring Response to Treatment of Metastatic Non-small Cell Lung Cancers
Brief Title: Early Assessment of Response to Treatment of Metastatic LUng Tumors Based on CIrculating Tumor DNA
Acronym: ELUCID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHD 160-18
Record Dates: First submitted 2019-04-16; First posted 2019-04-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ctDNA analysis (Experimental): additional blood sample of 20 ml
  Interventions: Other: ctDNA analysis

INTERVENTIONS:
Other: ctDNA analysis — blood sample at Baseline, 3weeks, 9 weeks after treatment, at progression if applicable

SUMMARY:
In patients with locally advanced or metastatic tumors, first-line therapeutic management is based on the use of targeted therapies (EGFR, BRAF ALK and ROS1 inhibitors), immunotherapies (anti-PD1/ anti-PDL1-antibodies or chemotherapy.

Despite patient selection based on histo-pathological and molecular criteria, not all patients respond to treatment. There are currently no markers to definitively guarantee a patient's response.

An alternative is to identify early patient response to treatment. The investigator hypothesize that change in circulating tumor DNA concentration (ctDNA) allow to early identify patients' therapeutic response (and non-response) of patients, regardless of the type of treatment used in the first line setting.

DETAILED DESCRIPTION:
The primary objective is to determine whether early evolution (between baseline and week 3) of circulating tumor DNA concentration predicts the radiological response to first-line treatment of advanced or metastatic NSCLC patients, regardless of treatment

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally advanced non-small cell lung cancer (stage III or IV)
* At least one measurable target according to RECIST criteria
* Identification of at least one molecular alteration in the tissue sample analyzed in the framework of patient management
* Performance Status 0 to 2
* Affiliated to a social security system
* Patient who can be followed under the protocol
* Patient agreed to participate in the study and gave his/her express consent

Exclusion Criteria:

* Minor
* Small cell or mixed bronchial cancer
* Radiotherapy (except radiotherapy for antalgic purposes) during the last 7 days
* Patient who has already started a first line of treatment
* Patient already included in an interventional research protocol that may have an impact on the results of the ELUCID study
* History of cancer (with the exception of non-melanoma skin, cervical cancer in situ, adequately treated) with sign of illness during the last 5 years
* Patient which, does present a substantial risk of recurrence.
* Major under guardianship, curators or deprived of liberty
* Pregnant or lactating woman, or of childbearing age without effective contraception
* Not affiliated to a social security system
* Inability to understand the protocol and / or to give express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Biological response at week 3 | week 3 after patient's recruitment date (baseline)
  Changes of the amount of ctDNA between baseline and week 3 will make it possible to determine the biological response: increase, stability or decrease in ctDNA.

SECONDARY OUTCOMES:
Progression-free survival (radiological assessment) and biological response at week 3. | week 3 after baseline
  Radiological assessment, based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria v1.1, will be: complete response, partial response, progression or stabilization. Biological response will be: increase, stability or decrease in ctDNA.
biological progression and radiological progression | progression
  Biological progression will be: increase in ctDNA - Radiological progression will be defined according to RECIST criteria v1.1 will be: progression
biological response and radiological response | progression
  Biological response will be: increase, stability or decrease in ctDNA and Radiological response will be defined according to RECIST criteria v1.1 will be: complete or partial response
Biological response and progression-free survival (radiological assessment) according to the therapeutic management: targeted therapies, immunotherapy, chemotherapy | week 3 after baseline
  Radiological assessment, based on RECIST criteria v1.1, will be: complete response or partial response. Biological response will be: increase, stability or decrease in ctDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Marc DENIS, Principal Investigator — CHD Vendee
Locations (2):
- France (2):
  - Marie MARCQ, La Roche-sur-Yon
  - Jaafar BENNOUNA, Nantes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herbreteau G, Marcq M, Sauzay C, Carpentier M, Pierre-Noel E, Pons-Tostivint E, Vallee A, Theoleyre S, Bizieux A, Bennouna J, Denis MG. Absolute Quantification of Nucleotide Variants in Cell-Free DNA via Quantitative NGS: Clinical Application in Non-Small Cell Lung Cancer Patients. Cancers (Basel). 2025 Feb 25;17(5):783. doi: 10.3390/cancers17050783. PMID 40075630